CLINICAL TRIAL: NCT05475509
Title: The Effect of Virtual Reality on Some Physiological and Psychological Parameters in Patients Receiving Chemotherapy After Breast Surgery (Mastectomy)
Brief Title: The Effect of Virtual Reality on Psychological Parameters in Patients Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Vesile Eskici Ilgin, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: vesile25
Record Dates: First submitted 2022-06-23; First posted 2022-07-27 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Side Effect of Chemotherapy
Keywords: anxiety; pain; tension; oxygen saturation
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: The research will be carried out by applying an experimental research design with a control group, pre-test-post-test applied, repetitive measurement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality group (nature videos were watched by wearing virtual reality glasses) (Experimental): In the experimental group, saliva sample will be taken before chemotherapy, Personal Information Form, State Anxiety Scale and VAS pre-test questionnaires will be applied, pre-test questionnaires will be applied to measure vital signs, and then virtual reality glasses will be introduced to the patients and the duration will vary between 3-10 minutes for a total of 30 minutes. A saliva sample will be taken and a post-test will be applied, with virtual reality glasses, videos with music background, park, nature and seaside walks, underwater, museum trips, videos that the patient wants to watch and can change whenever they want. Each patient will be shown the same video.
  Interventions: Other: Virtually reality
- Control Group (No Intervention): Personal Information Form, State Anxiety Scale and VAS pre-test questionnaires will be applied to the patients who accepted to participate in the study, saliva sample will be taken from the control group before chemotherapy, vital signs measurements will be made and post-test questionnaires will be applied at the 30th minute of chemotherapy, vital signs measurements will be made and saliva sample will be taken.

INTERVENTIONS:
Other: Virtually reality — Before chemotherapy, saliva samples will be taken from the control group, Personal Information Form, State Anxiety Scale and Visual Analogue Scale (VAS) pre-test questionnaires will be applied to the patients who accepted to participate in the study, vital signs measurements will be made and post-test questionnaires will be applied at the 30th minute of chemotherapy, vital signs measurements will be made, and A saliva sample will be taken. In the experimental group, a saliva sample will be taken before chemotherapy.
  Other Names: experimental-control group
  Arms: virtual reality group (nature videos were watched by wearing virtual reality glasses)

SUMMARY:
It has been determined that after mastectomy, women have psychological problems such as deterioration of body image, fear of losing their feminine characteristics and sexual dysfunction. Chemotherapy treatment for the first time causes patients to feel hopeless, to experience uncertainty and anxiety, and to increase their stress level. Experiencing intense stress during this treatment process can lead to severe mental problems, which negatively affects the course of the disease and the response to treatment. Chemotherapy is a painful procedure. Pain and stress are symptoms that affect each other positively.

Virtual reality glasses, which is one of the distraction methods used in the control of symptoms; It is widely used in clinical medical care to relieve symptoms by offering the possibility to create therapeutic environments in the evaluation and treatment of medical conditions. By affecting the emotional, cognitive, behavioral and sociocultural dimensions of the individual, it increases the sense of control, activity level and work capacity, reduces stress, pain, anxiety level, feeling of powerlessness and side effects of pharmacological methods.

DETAILED DESCRIPTION:
Breast cancer, which is common among women all over the world, draws attention in terms of mental and psychosocial aspects among cancer types because of the fear and anxiety of being cancer, as well as the loss of the breast, which appears as a symbol of femininity and sexuality, provides the nourishment of the baby, expresses love and motherhood feelings. type has been. Especially since it is a disease that evokes death, it creates more stress and anxiety in the individual compared to other diseases. In patients receiving chemotherapy after mastectomy, the side effects of the treatment, the treatment process, the fear of recurrence of the disease further increase the level of stress and anxiety. Nielsen, Zhang, Kristesen, and Schnohr, in their study examining the relationship between stress intensity and frequency, and breast cancer incidence, stated that women with high stress levels had a higher risk for breast cancer than women with low stress levels. Alacacioglu et al. The anxiety levels of female patients were found to be higher than male patients in their study with patients who were treated with chemotherapy. Karabulutlu et al., in their study with cancer patients, determined that 81.3% of cancer patients had depression and 61.5% had anxiety. In the study conducted by Aydoğan et al., the anxiety levels of cancer patients and healthy individuals were compared. found to be high. Non-pharmacological methods such as relaxation techniques, distraction, therapeutic touch, massage, hot-cold application, skin stimulation are used to reduce anxiety. In recent years, virtual reality as a distraction application has been widely used in clinical medical care to relieve pain. There are studies showing its effectiveness in pain and stress management in procedures such as injection applications, wound care, endoscopy procedure, phantom and chronic pain, chemotherapy applications. Schneider et al. During the chemotherapy treatment, videos were watched with virtual reality glasses to the patient with breast, lung and colon cancer who received chemotherapy treatment. It was determined that the anxiety and fatigue levels of the patients in the experimental group decreased and the time passed faster during the treatment process. Espinoza et al. Parks and nature walks were watched with virtual reality glasses in half-hour sessions consisting of four sessions for one week in 33 patients aged 41-85 years who were hospitalized in the oncology service and received chemotherapy treatment for metastatic cancer. After the application of virtual reality glasses, it was observed that the anxiety and depression levels of the patients decreased and the level of happiness increased.

According to the researchers' hypotheses, virtual reality acts as a non-pharmacological method, using cognitive and attentional processes on the body's complex pain modulation system. Although its neurobiological mechanisms have not been fully elucidated, studies have interestingly reported positive results in pain management. When patients feel that they are in the image, their attention is effectively distracted from the pain. Thus, the perception of pain is reduced. At the same time, distraction technique increases the patient's tolerance to pain, raises the pain threshold and causes him to feel less pain. This method, which is one of the independent practices of the nurse; It is a method frequently used in the current literature, as it is not an invasive procedure, is reliable, and has no known side effects. Although virtual reality is a potential and important technology in reducing the stress, pain and anxiety experienced during chemotherapy after mastectomy, there are limited or insufficient number of studies on this subject in our country. In the study of Toru, it was determined that virtual reality glasses applied during chemotherapy treatment in breast cancer patients reduced anxiety. In Karaman's study to determine the effect of virtual reality application on pain and anxiety during breast biopsy, found that virtual reality is effective on pain and anxiety.

However, unlike the studies conducted in this study, the stress level will be examined with saliva analysis and its relations with other parameters will be evaluated. There is no study directly related to this subject and it has been seen that a comprehensive study is needed. This research will be carried out to determine the effect of virtual reality on some physiological and psychological parameters in patients receiving chemotherapy after breast surgery. It is thought that the result of the research will contribute to the literature as an evidence-based non-pharmacological method in reducing the stress, pain and anxiety experienced during chemotherapy after mastectomy.

ELIGIBILITY:
Inclusion Criteria:

.Female patients who have had a mastectomy and will receive the first cure of outpatient chemotherapy

* Those between the ages of 18-75
* Willingness to participate in the research
* Absence of mental and communication problems
* No vision or hearing perception problem

Exclusion Criteria: • Under 18 and over 75 years old

* Patients who stopped participating in the study
* Patients with mental and communication problems

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The female gender was chosen because breast cancer is mostly seen in women.
Enrollment: 60 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS): | up to 24 hours
  VAS; It consists of a 10 cm long line starting with absence of pain (0) and ending with excruciating pain (10). The patient marks the severity of his pain on this line where he sees fit, this scale aims to explain the patient's pain in numbers.
Determination of Cortisol Level in Saliva: | up to 24 hours
  The UPLC-MS/MS system will be used for the determination of cortisol in saliva. A reverse phase C18 column will be used for the determination of cortisol. A mixture of 5 mM ammonium acetate and methanol (25: 75, v/v) will be used as the mobile phase. The flow rate will be determined as 0.25 ml/min. The injection volume will be 5 µL and the column oven temperature will be 25 °C. In analyzes performed in MRM mode, 363.2→121.1 ions will be selected.
State-Trait Anxiety Inventory (STAI I-II): | up to 24 hours
  The State-Trait Anxiety Inventory measures anxiety in adolescents over the age of 14 and adults. The scale, which is a type of self-assessment, includes 40 items consisting of short statements. 1-20 on the scale. questions, the state anxiety level of the individual, 21-40. The questions determine the level of trait anxiety. The total point value obtained from the inventory can vary between 20 and 80. A high score indicates a high level of anxiety, while a small score indicates a low level of anxiety.
Application Registration Form: | Investigators evaluate the change before and after chemotherapy in the 24-hour time frame.
  Pulse and oxygen saturation measurements of the patients before and after chemotherapy will be recorded in this form.

CONTACTS AND LOCATIONS:
Overall Officials: Vesile Eskici İlgin, PhD, Principal Investigator — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Palandöken, Turkey (Türkiye)